CLINICAL TRIAL: NCT02265835
Title: Anastomotic Airway Complications After Lung Transplantation : Risk Factors, Treatment Modalities and Outcome : a Single Center Experience.
Brief Title: Anastomotic Airway Complications After Lung Transplantation
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Yserbyt Jonas, MD, KU Leuven
Other Study IDs: ML6736
Record Dates: First submitted 2014-10-07; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Lung Transplantation; Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases of anastomotic airway complication: Cases of anastomotic airway complication
  Interventions: Other: no intervention
- Patients with normal anastomotic healing: Patients with normal anastomotic healing
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Retrospective analysis of data concerning anastomotic airway complications after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplantation

Exclusion Criteria:

* heart and lung transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung transplant recipients between 1/2005 en 12/2012
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
presence of anastomotic airway complication | 18 months
  Based upon radiological and endoscopic reports the presence and severity of anastomotic airway complications will be assessed.